CLINICAL TRIAL: NCT06084338
Title: Phase II Trial of Targeted Radiation With no Castration for Mcrpc
Brief Title: Randomized Phase II Trial of Targeted Radiation With no Castration for Mcrpc
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPLP-002-23M; 1I01CX002775 (NIH)
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: metastatic castration resistant prostate cancer; mCRPC; SBRT; Metastasis Directed Therapy; Lu177 PSMA; stereotactic body radiotherapy; stereotactic ablative radiotherapy; Pluvicto
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Metastasis directed therapy with stereotactic ablative radiotherapy to all detectable sites of disease plus PSMA radiopharmaceutical therapy and discontinuation of castration
  Interventions: Radiation: stereotactic ablative radiotherapy; Drug: Pluvicto
- Arm 2 (Experimental): Metastasis directed therapy with stereotactic ablative radiotherapy to all detectable sites of disease plus PSMA radiopharmaceutical therapy and discontinuation of castration, followed by restoration of physiologic testosterone
  Interventions: Radiation: stereotactic ablative radiotherapy; Drug: Pluvicto; Drug: topical testosterone

INTERVENTIONS:
Radiation: stereotactic ablative radiotherapy — Metastasis directed
  Other Names: SBRT
Drug: Pluvicto — PSMA targeted radiopharmaceutical therapy
  Other Names: Lu177-PSMA
Drug: topical testosterone — Topical testosterone 1.62% gel
  Other Names: androgel
  Arms: Arm 2

SUMMARY:
This trial tests if the combination of comprehensive metastasis directed therapy delivered by a precision form of external beam radiotherapy (stereotactic ablative radiotherapy), combined with PSMA targeted radiopharmaceutical therapy and cessation of castration, and then followed by testosterone replacement, is an effective treatment for metastatic castration resistant prostate cancer.

All patients will be treated with stereotactic ablative radiotherapy and PSMA targeted radiopharmaceutical therapy with cessation of castration. Half of patients are randomized to either receive, or not receive, subsequent testosterone replacement.

DETAILED DESCRIPTION:
This is a randomized, parallel-arm, two-stage open-label phase 2 study of comprehensive metastasis directed therapy in the form of stereotactic body radiation therapy (SBRT) to all detectable sites of disease plus PSMA targeted radiopharmaceutical therapy (pluvicto), discontinuation of castration, with and without testosterone replacement therapy (TRT) in metastatic castration resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older at the time the Informed Consent is signed
* The subject (or legally acceptable representative if applicable) must provide written informed consent for the trial
* Pathologic diagnosis of prostate cancer of adenocarcinoma histology; presence small cell/neuroendocrine carcinoma is exclusionary
* Metastatic disease as documented by:

  * Osseous metastases detected by technetium-99m (99mTc) planar bone scan or NaF PET scan, or CT scan at some point in patient's history
  * Soft tissue metastases documented on CT or MRI
* PSMA avid metastatic disease as determined by 18F-DCFPyL: at least one lesion with PSMA avidity greater than that of liver (see Prescribing Information for Pluvicto)
* Progressive castration resistant prostate cancer as defined by serum testosterone < 50 ng/mL and one of the following:

  * PSA progression confirmed per Prostate Cancer Clinical Trials Working Group (PCWG3)
  * Radiographic progression of soft tissues according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) modified based on PCWG3, or radiographic progression of bone according to PCWG3
* Prior use of a novel AR signaling inhibitor for 4 weeks, including abiraterone acetate plus prednisone/prednisolone, enzalutamide, apalutamide, and/or darolutamide

NOTE: These AR signaling inhibitors may have been used for mCSPC, M0CRPC, and/or mCRPC.

* ECOG PS grade of 0-2
* 10 metastases detectable on molecular imaging (PSMA and FDG PET) and amenable to SBRT

  * 20% of metastases that are FDG avid but PSMA negative
  * Metastases that are not detectable on PSMA and FDG PET do not count toward the total number of metastases, as they are presumed to represent adequately treated sites of disease
* Life expectancy 6 months
* Adequate organ function:

  * Hemoglobin (hgb) > 8.0 g/dL
  * Absolute neutrophil count (ANC) > 1500/ µL
  * Platelets > 75,000/ µL
  * Total bilirubin 1.5 x ULN OR direct bilirubin ULN for participants with total bilirubin levels >1.5 x ULN
  * ALT and AST 3.0 x ULN ( 5 x ULN for participants with liver metastases) (Child-Pugh class A and B allowed; Child-Pugh class C is excluded)
  * Creatinine < (2.0 mg/dL) during screening evaluation (>2.0 is allowed if EGFR >30 mL/min/1.73 m2)
* Subject must agree to use contraception during the treatment period plus an additional 120 days after the last dose of study treatment and must refrain from donating sperm during this period

Exclusion Criteria:

* Visceral metastases including liver and brain (lung metastases are allowed)
* Small cell/neuroendocrine carcinoma by hematoxylin and eosin light histology (immunohistochemical detection of rare/occasional cells that stain for neuroendocrine markers such as synaptophysin, neuron specific enolase, or chromogranin A is not sufficient to make a diagnosis of small cell/neuroendocrine carcinoma)
* Anti-neoplastic therapies for prostate cancer must be completed > 2 weeks prior to Day 1 (initiation of first dose of PSMA RLT)

  * Investigational agents must have been completed > 4 weeks of Day 1

Note: Participants must have recovered from all AEs due to previous therapies to Grade 1 or baseline

* Participants with Grade 2 neuropathy may be eligible

  * Herbal and non-herbal products that may decrease PSA levels other than medical castration and megestrol (up to 40 mg/day is allowed) for hot flashes
  * Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* If a subject has undergone major surgery, they must have recovered adequately from the toxicities or complications from the intervention within 4 weeks prior to starting therapy
* History of non-prostate active malignancy requiring treatment in the 24 months prior to Day 1 except for non-muscle invasive urothelial cancer, non-melanoma skin cancer, or any cancer that in the opinion of the investigator has been adequately treated and will not interfere with study procedures or interpretation of results
* Active infection or conditions requiring treatment with antibiotics
* Symptomatic local recurrence in the setting of prior curative intent therapy (surgery and/or radiation to the prostate)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Subject is planning to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Current or impending cord compression or another indication for urgent palliative radiation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient must have or have had a prostate
Enrollment: 60 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month radiographic progression-free survival (rPFS) | 6-months
  6-month radiographic progression-free survival (rPFS) measured by conventional imaging from date of initiation of PSMA radiopharmaceutical therapy

SECONDARY OUTCOMES:
safety as assessed by physician reported toxicity | up to two years
  Physician reported Common Terminology Criteria for Adverse Events (CTCAE version 5.0)
Patient reported health-related quality of life measured by Expanded Prostate Cancer Index Composite (EPIC-26) | up to two years
  EPIC-26 contains 26 items in 5 domains (Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal). Raw scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
PSA30, PSA50, PSA90, maximal PSA response | up to two years
  This is the rate of PSA response (PSA decrease by 30%, 50%, 90%), and maximal response
Time to PSA progression | up to two years
  Time to PSA progression per PCWG3 criteria, from date of initiation of PSMA radiopharmaceutical therapy
Objective response rate | up to two years
  Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) from date of initiation of PSMA radiopharmaceutical therapy
Time to radiographic progression | up to two years
  Time-to-event, Bone progression by Prostate Cancer Working Group 3 (PCWG3) criteria and/or soft tissue progression by RECIST v1.1, from date of initiation of PSMA radiopharmaceutical therapy
PSMA PET response | up to two years
  Measured using Prostate Cancer Molecular Imaging Standardized Evaluation (PROMISE)
Progression Free Survival | up to two years
  Time-to-event, a composite between time to PSA progression (PCWG3) and/or radiographic progression (PCWG3 for bone, RECIST 1.1 for soft tissue), from date of initiation of PSMA radiopharmaceutical therapy
Overall survival | up to two years
  Time-to-event, from date of initiation of PSMA radiopharmaceutical therapy
Patient reported health-related quality of life measured by The Functional Assessment of Cancer Therapy-Prostate (FACT-P). | up to two years
  FACT-P includes a general functional status scale (consisting of four subscales: physical wellbeing, social and family wellbeing, emotional wellbeing, and functional wellbeing) and a prostate-cancer-specific subscale. Total score is calculated with general function and prostate-cancer-specific scores, and ranges from 0 to 156 (higher scores indicate better functional status).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas George Nickols, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (4):
- United States (4):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No